CLINICAL TRIAL: NCT01349478
Title: Electrical Stimulation Induced Lower Limb Exercise Capacity, Cardiorespiratory Response, Cardiovascular Risk Factors and Muscle Activity Patterns in Response to Robotic Assisted Treadmill Gait Training in Individuals With Complete Motor Spinal Cord Injury
Brief Title: The Effects of Passive Gait Training in Complete Motor Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Gabriel Zeilig (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Gabriel Zeilig, Dr. Gabriel Zeilig, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHEBA-11-8422-GZ-CTIL
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Motor Complete Spinal Cord Injury
Keywords: paraplegia; tetraplegia; passive gait training; O2 consumption; exercise capacity; CVD risk factors; spasticity; pain; bladder, bowel; well being
MeSH Terms: conditions — Paraplegia; Quadriplegia; Muscle Spasticity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental)
  Interventions: Device: LOKOMAT

INTERVENTIONS:
Device: LOKOMAT — Robot-assisted gait training,8 weeks,3 sessions a week,20-45 min each session.
  Other Names: driven gait orthosis

SUMMARY:
The purpose of this study is to determine whether a three times per week, 2 month robotic assisted treadmill gait training program, will beneficially affect the fitness, physical and psychological well-being, and the vascular and metabolic cardiovascular risk factors in individuals with complete motor Spinal Cord Injury (SCI).

DETAILED DESCRIPTION:
Cardiovascular morbidity and mortality are a source of increasing concern among people with SCI and their health providers. The importance of physical activity in reducing the risk of heart disease in this population is indisputable, but exercise opportunities for persons with SCI are limited by physiologic and functional factors. Decreased functional muscle mass, impaired autonomic control of myocardial function, and decreased venous return limits training responses.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant non-lactating female
* At least 6 months after injury
* Complete (AIS A-B) cervical (C4-8) or thoracic (T1-T6) spinal cord injury according to American Spinal Injury Association (AIS) guidelines.
* Under 100 kg and between 155 - 200 cm of height

Exclusion Criteria:

* History of severe neurological injuries other than SCI (MS, CP, ALS, TBI etc).
* Severe concurrent medical diseases: infections, heart or lung, pressure sores, etc
* Unstable spine or unhealed limbs or pelvic fractures
* Psychiatric or cognitive situations that may interfere with the trial
* Spasticity above 3 degree according to Ashworth scale
* Reduced range of motion of knee/hip > 15°

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Electrical stimulation induced lower limb exercise capacity in individuals with SCI | 4 and 8 weeks of training
  The lower limb exercise capacity in response to electrical stimulation will be measured by the use of the ERGYS II system

SECONDARY OUTCOMES:
Reduction of risk factors for CVD | 4 and 8 weeks
  1. Plasms levels of: Total cholesterol, LDL-C, HDL-C, TC/HDL, LDL/HDL, CRP, Triglycerides, IL6, fasting glucose and fasting insulin
  2. blood pressure, O2 consumption, CO2 production, O2 saturation, Heart rate, RER max (respiratory exchange ratio), VE (minute ventilation), AT (Anaerobic Threshold), Work rate max

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Zeilig, M.D, Principal Investigator — Sheba Medical Center; Moshe Berg, Medical Student, Study Director — Sheba Medical Center; Evgeni gaidukov, M.D, Study Director — Sheba Medical Center; Shirley Ackerman-Laufer, B.A, Study Director — Sheba Medical Center; Shlomit Siman, B.A., Study Director — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel

REFERENCES:
- [Background] American Spinal Injury Association/International Medical Society of Paraplegia International Standards for Neurological and Functional Classification of Spinal Cord Injury Patients. Chicago, IL: American Spinal Injury Association/International Medical Society of Paraplegia; 2000.
- [Background] Marino RJ Reference Manual American Spinal Cord Association 2000
- [Background] Lucin KM, Sanders VM, Jones TB, Malarkey WB, Popovich PG. Impaired antibody synthesis after spinal cord injury is level dependent and is due to sympathetic nervous system dysregulation. Exp Neurol. 2007 Sep;207(1):75-84. doi: 10.1016/j.expneurol.2007.05.019. Epub 2007 Jun 2. PMID 17597612
- [Background] Bauman WA, Spungen AM, Adkins RH, Kemp BJ. Metabolic and endocrine changes in persons aging with spinal cord injury. Assist Technol. 1999;11(2):88-96. doi: 10.1080/10400435.1999.10131993. PMID 11010069
- [Background] De Vivo MJ Long term survival and causes of death in Spinal Cord Injury Clinical Outcomes from the model systems 1995
- [Background] Svircev JN. Cardiovascular disease in persons with spinal cord dysfunction-an update on select topics. Phys Med Rehabil Clin N Am. 2009 Nov;20(4):737-47. doi: 10.1016/j.pmr.2009.06.012. PMID 19781509
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Teasell RW, Arnold JM, Krassioukov A, Delaney GA. Cardiovascular consequences of loss of supraspinal control of the sympathetic nervous system after spinal cord injury. Arch Phys Med Rehabil. 2000 Apr;81(4):506-16. doi: 10.1053/mr.2000.3848. PMID 10768544
- [Background] Jacobs PL, Nash MS. Exercise recommendations for individuals with spinal cord injury. Sports Med. 2004;34(11):727-51. doi: 10.2165/00007256-200434110-00003. PMID 15456347
- [Background] Bhambhani YN, Eriksson P, Steadward RD. Reliability of peak physiological responses during wheelchair ergometry in persons with spinal cord injury. Arch Phys Med Rehabil. 1991 Jul;72(8):559-62. PMID 2059132
- [Background] Pollack SF, Axen K, Spielholz N, Levin N, Haas F, Ragnarsson KT. Aerobic training effects of electrically induced lower extremity exercises in spinal cord injured people. Arch Phys Med Rehabil. 1989 Mar;70(3):214-9. PMID 2784311
- [Background] Israel JF, Campbell DD, Kahn JH, Hornby TG. Metabolic costs and muscle activity patterns during robotic- and therapist-assisted treadmill walking in individuals with incomplete spinal cord injury. Phys Ther. 2006 Nov;86(11):1466-78. doi: 10.2522/ptj.20050266. PMID 17079746
- [Background] Hidler J, Hamm LF, Lichy A, Groah SL. Automating activity-based interventions: the role of robotics. J Rehabil Res Dev. 2008;45(2):337-44. doi: 10.1682/jrrd.2007.01.0020. PMID 18566951
- [Background] Hutchinson KJ, Gomez-Pinilla F, Crowe MJ, Ying Z, Basso DM. Three exercise paradigms differentially improve sensory recovery after spinal cord contusion in rats. Brain. 2004 Jun;127(Pt 6):1403-14. doi: 10.1093/brain/awh160. Epub 2004 Apr 6. PMID 15069022
- [Background] Thoumie P, Le Claire G, Beillot J, Dassonville J, Chevalier T, Perrouin-Verbe B, Bedoiseau M, Busnel M, Cormerais A, Courtillon A, et al. Restoration of functional gait in paraplegic patients with the RGO-II hybrid orthosis. A multicenter controlled study. II: Physiological evaluation. Paraplegia. 1995 Nov;33(11):654-9. doi: 10.1038/sc.1995.137. PMID 8584300
- [Background] Eng JJ, Levins SM, Townson AF, Mah-Jones D, Bremner J, Huston G. Use of prolonged standing for individuals with spinal cord injuries. Phys Ther. 2001 Aug;81(8):1392-9. doi: 10.1093/ptj/81.8.1392. PMID 11509069
- [Background] Mark S. Nash. Cardiovascular Fitness and Exercise Prescription after Spinal Cord Injury. Spinal Cord Medicine. Principles and Practice. Vernon W. Lin 2010 pages 848-855